CLINICAL TRIAL: NCT00004475
Title: Molecular Genetics of Hereditary Pancreatitis
Brief Title: Genetic Linkage Study for Hereditary Pancreatitis
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Whitcomb, Principal Investigator, University of Pittsburgh
Other Study IDs: PRO07090243
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or saliva samples are collected from patients and family members. DNA is extracted and used for genotypic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to establish linkage in families with hereditary pancreatitis (HP) to the cationic trypsinogen gene or other, as yet unknown, HP gene(s).

DETAILED DESCRIPTION:
Hereditary Pancreatitis (HP) is an inflammatory condition of the pancreas which is usually recurrent in nature and occurs in blood-related persons over two or more generations. It is an autosomal dominant trait with complete penetrance by variable expression. Symptoms are usually present during childhood and it is the second most common cause of chronic or recurrent pancreatitis in children. HP is a primary disorder and can therefore be differentiated from other inherited disorders that cause secondary pancreatitis. The purpose of this study is to establish linkage in families with HP between the phenotype and a chromosomal locus (loci) which contains the responsible gene. Affected families are recruited to donate a blood sample through referral from their primary physician or self-referral. The potential significance lies in the identification of the genetic defect causing HP and understanding the pathophysiologic mechanism of the disease. Typically families with HP have a high incidence of adenocarcinoma of the pancreas and identification of the cause of this disease may provide critical insights into the cause of pancreatic cancer.

Blood samples are collected from patients and family members. DNA is extracted from the blood and used for genotypic analysis and linkage analysis. Patients do not necessarily receive the results of the genetic testing and the results do not influence the type or duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pancreatitis at age < 60 OR
2. Diagnosis of pancreatitis at any age and at least one other 1st or 2nd degree relative with a diagnosis of pancreatitis or pancreatic cancer OR
3. Diagnosis of pancreatic cancer and a 1st or 2nd degree relative with pancreatic cancer or pancreatitis OR
4. Diagnosis of pancreatic insufficiency or maldigestion that improves with pancreatic enzyme replacement OR
5. Close family members (parents, grandparents, siblings cousins - anyone related by blood) of subjects who meet criteria 1, 2, or 3 AND
6. Age 3 months up to 100 years

Exclusion Criteria:

There are no general exclusions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Diagnosis of hereditary pancreatitis with confirmation of phenotype by: Onset of pain before age 20 Amylase elevation at least 2 times normal Surgical or postmortem confirmation of pancreatitis Unequivocal evidence of pancreatic exocrine insufficiency in the absence of trauma, alcohol abuse, elevated serum lipids, or other known causes
  * Family member of a patient diagnosed with hereditary pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 808 (Actual)
Dates: Start 1998-12 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Whitcomb, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Presbyterian University Hospital, Pittsburgh, Pennsylvania, United States